CLINICAL TRIAL: NCT03352947
Title: INTERIM: a Randomised Phase II Feasibility Study of INTERmittent Versus Continuous Dosing or Oral Targeted Combination Therapy in Patients With BRAFV600 Mutant Stage 3 Unresectable or Metastatic Melanoma
Brief Title: Continuous vs Intermittent Dabrafenib Plus Trametinib in BRAFV600 Mutant Stage 3 Unresectable or Metastatic Melanoma
Acronym: INTERIM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Oxford University Hospitals NHS Trust (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, CCTU- Cancer Theme, Consultant and Associate Lecturer in Medical Oncology, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INTERIM; 2016-005228-27 (EudraCT Number); PB-PG-0815-20048 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2017-11-09; First posted 2017-11-24 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Intervention Model Description: INTERIM is a multi-centre, open label, two arm, randomised phase II feasibility trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous (Standard) (Active Comparator): Dabrafenib 150mg twice daily 12 hours apart, on days 1-28 of a 28 day cycle plus Trametinib 2mg once daily, on days 1-28 of a 28 day cycle
  Interventions: Drug: Dabrafenib; Drug: Trametinib
- Intermittent (experimental) (Experimental): Dabrafenib 150mg twice daily 12 hours apart, on days 1-21 of a 28 day cycle plus Trametinib 2mg once daily, on days 1-14 of a 28 day cycle
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — 150mg Dabrafenib twice daily day 1-21 of 28 day cycle in intermittent arm Day 1-28 of 28 day cycle in continuous arm
  Other Names: Tafinlar
Drug: Trametinib — Trametinib 2mg once daily Day 1-14 of a 28 day cycle in intermittent arm Day 1-28 of a 28 day cycle in the continuous arm
  Other Names: Mekinist

SUMMARY:
This feasibility study aims to determine if intermittent dosing is deliverable, based on patient and professional willingness to take part in a randomised trial evaluating less rather than the standard durations of treatment. The trial will evaluate treatment compliance, Progression Free Survival and Quality of Life, to inform whether a subsequent definitive trial is justified and how it should be designed.

DETAILED DESCRIPTION:
Metastatic melanoma has a very poor prognosis: median overall survival is 8 months untreated and around 2 years even with optimal systemic therapies. A gene called BRAF is abnormal in about half of melanomas and biological agents targeting the BRAF pathway have been shown to extend life. They are now routinely available in NHS clinical practice.

Giving BRAF and MEK inhibitor drugs together offers the best anti-cancer treatment for these patients. However, treatment is limited by side-effects (often affecting the skin) and secondary resistance (which means the cancer regrows usually after about a year).

Laboratory experiments and case reports suggest intermittent dosing of these chronic orally administered drugs makes BRAF pathway inhibitors work for longer, extending life and reducing side effects. The INTERIM trial aims to test whether less treatment than usual is acceptable to patients and doctors and, potentially, more beneficial. The INTERIM trial also aims to develop better tools to monitor skin side-effects.

The target population will be male and female participants aged 18 and over with BRAFV600 mutant stage 3 unresectable or metastatic melanoma.Patients will be provided with information regarding the trial both through conversation with investigators and research nurses and in writing via a patient information sheet. Patients will be given time to ask questions and discuss with family/support structures before deciding to participate. If the patient agrees to take part, they will be asked to provide written consent.

Visit schedule for consenting patients:

Screening:

Consenting patients will enter the screening/baseline phase, which will be completed within 28 days prior to randomisation. This will include assessing the patient against inclusion & exclusion criteria.

Randomisation:

If eligible, patients will be randomly assigned to either treatment arms using a web-based central randomisation system. Patients will be randomised on a 1:1 basis to one of 2 arms:

Control arm: dabrafenib 150mg twice daily and trametinib 2mg once daily, taken by mouth continuously on a 4 week cycle Experimental arm: dabrafenib 150mg twice daily x 3 weeks and trametinib 2mg once daily x 2 weeks, on a 4 week cycle

On treatment:

During the first two cycles of treatment patients will attend the hospital every two weeks (on days 1 and 15 of the cycle) where they will have a clinical review.

From cycle 3 onwards patients will attend the hospital only on day 1 of the cycle.

If patients are on treatment for more than 52 weeks, clinic visits can be every other cycle with telephone follow-up between to ensure patient review is at least every 4 weeks until progression.

End of Treatment:

At the end of treatment an additional clinical visit will be performed to review the patient. If at the time of treatment cessation patients have not met the criteria for disease progression they will be followed up every 4 weeks. After 52 weeks since randomisation there will be the option of clinic visits every 8 weeks with telephone follow-up in between.

Disease progression:

Patients will have a clinical visit at the time of protocol-defined disease progression.

Follow-up after disease progression:

Patients will attend hospital every three months after disease progression for a minimum of 9 months from randomisation.

Trial procedures:

Clinical review & physical examinations:

Patients will be reviewed by the trial team during the screening period, at every treatment and follow-up visit. This will involve recording any medications they may be taking, and any symptoms and/or side-effects they may have. Patients will also have a physical examination, and assessment of blood pressure as part of this review, and the clinical team will assess the patient's clinical status using ECOG and Karnofsky performance status scales.

Baseline skin assessment & skin toxicity questionnaires:

At screening the patient and clinician will be asked to complete a questionnaire about the baseline condition of the patient's skin. If during treatment there are any skin-related adverse events both the patient and clinician will be asked to complete a skin toxicity questionnaire.

Compliance assessment:

During treatment at each clinical visit the patient will be asked to bring their medication along with their diary card.The clinical team will record how many tablets remain and how many tablets have been taken. The patient will be asked to record in the diary card the date and time when they take their medication. Both of these activities will be used to assess the patient's compliance to the treatment regimen.

Pregnancy test:

Women of child bearing potential will have a pregnancy test at screening to ensure they are not pregnant and are therefore able to receive the trial drugs.

Electrocardiogram (ECG):

An ECG test is required before starting the trial.

Echocardiogram (ECHO):

An ECHO is required prior to starting the trial in patients with a history of cardiac problems, in patients with no cardiac history and a normal ECG it must be performed within two weeks of starting trial drug. ECHOs will subsequently be performed as standard of care, the recommended frequency is during cycle 4 and every 12 weeks thereafter to ensure that patients are tolerating the trial drugs well.

Blood samples (routine and research):

Patients will be asked to have routine blood tests (FBC, renal, liver, bone profiles, LDH) to ensure that they are fit enough for the trial, and that they are tolerating the drug well. These blood samples will be taken at every clinical visit during treatment and at disease progression.

Patients will also be asked to give extra blood for research related to this trial. The samples will be used to measure circulating tumour DNA (ctDNA). An extra blood sample will be taken every 2 weeks for the first two cycles of treatment, every 4 weeks for the next two cycles, then every 8 weeks, and at disease progression.

Patients will be asked if they wish to participate in optional pharmacokinetic sampling. This will involve collection of 9 blood samples on both cycle 1 day 1, and cycle 2 day 15 at timepoints after they have taken their tablets. Additionally, 3 blood samples would be taken if their disease progresses.

Tumour assessments:

Patients will have an initial CT scan of body and head during the screening period. Scans will be repeated between days 8-15 of cycle 2 and then every 8 weeks until the end of treatment. If treatment continues beyond 52 weeks imaging can be reduced to every 12 weeks. If the initial screening head scan is clear, the head scan only requires repeating at every other assessment.

Quality of Life questionnaires:

Patients will be asked to fill in questionnaires about their quality of life at screening on day 1 of cycle 2, and then every12 weeks until the end of participation in the trial.

Tumour Tissue collection:

Upon starting treatment patients will be asked to donate previously archived tissue collected for research purposes. If patients undergo surgical resection or biopsy during the course of the trial for progressive disease, a tumour sample will be requested for this research.

Patient Experience survey:

Patient who do not consent to participate in the trial will be asked to complete a questionnaire to explore their reasons for declining. Additionally, patients who do participate in the trial will be asked to complete patient experience questionnaires after consent and after 9 months participation in the trial. These questionnaires will ask the patients about their experience of participating in the trial and any toxicity they experienced.

Patients may continue on allocated treatment as long as they benefit from the treatment and it is tolerable. Patients will be followed for a minimum of 9 months from randomisation to a maximum of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥18 years old
* Histologically or cytologically confirmed BRAFV600 mutant stage 3 unresectable or metastatic melanoma
* Measurable disease by RECIST
* ECOG performance status 0-2
* Minimum life expectancy 12 weeks
* Adequate bone marrow, renal and liver function
* Received no prior BRAF or MEK inhibitor therapy for metastatic disease
* Willing and able to comply with the scheduled visits, treatment plans, laboratory tests, completion of QoL questionnaires and other study procedures
* Archival tumour tissue sample available
* Women of child-bearing potential and all sexually active male patients must agree to use effective contraception methods throughout treatment

Exclusion Criteria:

* Concomitant immunotherapy being administered to treat advanced melanoma
* Other invasive malignancies diagnosed within the last year which are not in complete remission, or for which additional therapy is required
* Significant acute or chronic medical or psychiatric condition, disease or laboratory abnormality which in the judgment of the investigator would place the patient at undue risk or interfere with the trial
* Women who are pregnant, plan to become pregnant or are lactating during the trial period
* Other investigational anti-cancer drugs
* Use of strong inducers and inhibitors of CYP3A or CYP2C8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | To be assessed once the trial has been recruiting for 15 months, or when 15 sites have been open for 6 months whichever is sooner
  Average number of patients recruited per site per two months.
Treatment compliance | 6 months from randomisation
  percentage of patients completing the allocated treatment
Overall Quality of Life | 6 months from randomisation
  global health status score derived from (EORTC) QLQ-C30 questionnaire
Progression Free survival | calculated as the duration from the date of randomisation to the date of first progression or death from any cause, whichever occurs first, assessed up to 5 years
  Assessed according to standard Response Criteria in Solid Tumours (RECIST v1.1)

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events (safety and tolerability) | Through study completion, an average of 1 year
  Assess using standard cancer National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) V4.03)
Objective response rate | Through study completion, an average of 1 year
  assessed according to RECIST v1.1
Time to treatment failure | Through study completion, an average of 1 year
  Time from starting drug treatment (day 1, cycle 1) until day 1 of last cycle + 28 days
Overall survival | Assessed up to 5 years
  calculated as duration from date of randomisation to the date of death from any cause
Patient Reported Outcomes focusing on skin toxicity evaluation | Through study completion, an average of 1 year
  assessed using skin-specific patient reported outcome measures
Patient Experience | Surveys at screening and after 9 months. Interviews by invitation at a later date
  Surveys of patients in both arms of the trial. Semi-structured interview in a subset of patients.
Impact on Quality of Life | At 6 months from baseline
  Using EORTC QLQ-C30 questionnaire
Health Economic Evaluation | Through study completion, an average of 1 year
  Using EQ-5D 5L questionnaire

OTHER OUTCOMES:
Kinetics of BRAF mutation load in each arm of the trial | Through study completion, an average of 1 year
  using blood and tumour tissue taken from recruited patients
Emerging genetic changes associated with acquired resistance | Through study completion, an average of 1 year
  using blood and tumour tissue taken from recruited patients

CONTACTS AND LOCATIONS:
Overall Officials: Pippa Corrie, FRCP, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No
PID will not be shared with other researchers. PID will not be moved from participating sties. Patient will be identified by their initials, date of birth and trial number.

DOCUMENTS (1):
  • Study Protocol (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT03352947/Prot_000.pdf